CLINICAL TRIAL: NCT00038233
Title: Thalidomide for Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM98-359
Record Dates: First submitted 2002-05-29; First posted 2002-05-30 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Multiple Myeloma
Keywords: myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thalidomide (Experimental): 200 mg at bedtime daily for 14 days (days 1-14), followed by an increase to 400 mg daily for 14 days (days 15-28), 600 mg daily for 14 days (days 29-42), up to a maximum 800 mg (days 43-completion)
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — 200 mg at bedtime daily for 14 days (days 1-14), followed by an increase to 400 mg daily for 14 days (days 15-28), 600 mg daily for 14 days (days 29-42), up to a maximum 800 mg (days 43-completion)
  Other Names: Thalomid

SUMMARY:
The objective of this protocol is to assess therapeutic activity of thalidomide in previously untreated patients with asymptomatic multiple myeloma.

DETAILED DESCRIPTION:
This study attempts to examine the potential efficacy of thalidomide in the treatment of patients with previously untreated multiple myeloma. The trial focuses on patients with asymptomatic and indolent disease who do not require immediate chemotherapy. We intend to treat asymptomatic patients with an initial dose of 200 mg each evening, increasing to a maximum of 800 mg.

Thalidomide is supplied as 50 mg capsules to be taken by mouth. The initial dose will be 200 mg at bedtime daily for 14 days (days 1-14), followed by an increase to 400 mg daily for 14 days (days 15-28), 600 mg daily for 14 days (days 29-42), up to a maximum 800 mg (days 43-completion) daily provided there are no side effects.

Patients who experience significant toxicity (grade 2 or more) at any time during therapy will receive a lower dose after treatment is interrupted for at least 2 days.

Once a maximum tolerated dose has been reached free of side effects, that dose will be continued for a total of 3 months from institution of therapy before definition of response or resistance. Only patients who have received at least 200 mg/d for at least 2 months will be considered evaluable for response. For patients in remission, treatment will be continued at the maximum dose free of side effects until relapse. Selected patients <55 years of age who achieve remission may be eligible for stem cell transplant (SCT) in which case thalidomide will be discontinued prior to SCT.

Patients must be willing to return for evaluation every 4 weeks since thalidomide may only be prescribed for 28 day intervals.

ELIGIBILITY:
* Previously untreated patients with multiple myeloma and without serious or imminent complications (e.g. impending pathologic fracture, hypercalcemia, renal insufficiency). All asymptomatic patients with low or intermediate tumor mass will qualify.
* Patients with high tumor mass, symptomatic or impending fractures, hypercalcemia (corrected calcium >11.5 mg%), anemia (Hgb <8.5 gm/dl), renal failure (creatinine >2.0 mg/dl), high serum lactate dehydrogenase (>300 U/L) or plasma cell leukemia (>1000/ul) are ineligible.
* Overt infections or unexplained fever should be resolved before treatment. Adequate liver function (including SGPT, bilirubin and LDH) is required.
* Patients must have Zubrod performance of 1 or less.
* Patients must provide written informed consent indicating that they are aware of the investigational nature of this study.
* Life expectancy should exceed 1 year.
* Patients with idiopathic monoclonal gammopathy and non-secretory multiple myeloma are ineligible. Patients whose only prior therapy has been with local radiotherapy, alpha-IFN, or ATRA are eligible. Patients exposed to prior high-dose glucocorticoid or alkylating agent are not eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 1999-05; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of Thalidomide | 14 day cycles

CONTACTS AND LOCATIONS:
Overall Officials: Donna M. Weber, MD, BS, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org